CLINICAL TRIAL: NCT07278674
Title: Clinical Study of Eflornithine After Immunotherapy for High-risk Neuroblastoma（CSHEIN）
Acronym: CSHEIN
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Children's Hospital (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiChildrens
Record Dates: First submitted 2025-02-08; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: High Risk Neuroblastoma
Keywords: High risk neuroblastoma; Eflornithine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Oral administration of eflornithine for the prevention of high-risk neuroblastoma — This study is a single arm clinical observational study and does not involve control interventions
  Other Names: No other intervention measures

SUMMARY:
Evaluate the impact of maintenance therapy with eflornithine on event-free survival and overall survival in high-risk neuroblastoma (NB) children after immunotherapy, and assess its safety.

DETAILED DESCRIPTION:
The investigators plan to recruit 20 participants and divide them into Group A and Group B based on their clinical status. The inclusion criteria for Group A are: newly diagnosed high-risk neuroblastoma (NB) patients who have completed the standard treatment plan (including immunotherapy) and whose disease has reached complete response (CR) or very good partial response (VGPR). The inclusion criteria for Group B are: recurrent or refractory NB patients who have completed any treatment for recurrent disease, or who have achieved disease stability after any salvage or intensification therapy for primary refractory disease, with at least a partial response (PR) as assessed by CT or MRI and negative bone marrow aspiration. There are no restrictions regarding gender or geographic region. Participants must be under 18 years of age. Eligible subjects will be enrolled into the study after receiving the first oral dose of eflornithine, with a total treatment course of 2 years. Follow-up will continue for up to 3 years after completion of eflornithine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. According to the International Neuroblastoma Risk Group Classification, it has been histologically diagnosed as high-risk NB.
2. Under the age of 18.
3. The disease assessment status is PR (via CT or MRI) and the bone marrow smear is negative.
4. If the residual mass is MIBG negative or MIBG positive and lacks FDG-PET affinity, it is considered evidence that the mass does not represent active disease. Subjects with stable residual tumor mass visible on CT/MRI will be included in the study.
5. Qualified hematological parameters and organ function; Refer to the CI CTC 4.0 adverse reaction grading standard of grade 2 and below.
6. Eflornithine needs to be activated within 120 days after the completion of previous treatment.

Exclusion Criteria:

1. According to the International Neuroblastoma Risk Group Classification, it has been histologically diagnosed as non high risk NB.
2. Prior to enrollment, the disease assessment status was either progressive disease (PD) or relapse (via CT or MRI).
3. Positive bone marrow smear.
4. Hematological parameters and organ function are not qualified, according to the CI CTC 4.0 adverse reaction grading standard of grade 3 or above.
5. The guardian does not agree to participate.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with high-risk neuroblastoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
The event free survival rate after the completion of the first DFMO | 5 years
  The event free survival rate of high-risk NB patients who complete standard treatment and take oral eflornithine after immunotherapy.
overall survival rate after the completion of the first DFMO | 5 years
  overall survival rate of high-risk NB patients who complete standard treatment and take oral eflornithine after immunotherapy.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 5 years
  This study will comprehensively evaluate the safety and tolerability of eflornithine. The primary assessments include the incidence and severity of all treatment-emergent adverse events (graded per NCI CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Jingbo Shao, PhD，chief physician, Principal Investigator — Shanghai Children's Hospital; Wen Su, PhD，associate chief physician, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Hainan Branch, affiliated with Shanghai Jiao Tong University School of Medicine and Children's Hospital of Shanghai, affiliated with Shanghai Jiao Tong University School of Medicine, Hainan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duke ES, Bradford D, Sinha AK, Mishra-Kalyani PS, Lerro CC, Rivera D, Wearne E, Miller CP, Leighton J, Sabit H, Zhao H, Lane A, Scepura B, Pazdur R, Singh H, Kluetz PG, Donoghue M, Drezner N. US Food and Drug Administration Approval Summary: Eflornithine for High-Risk Neuroblastoma After Prior Multiagent, Multimodality Therapy. J Clin Oncol. 2024 Sep 1;42(25):3047-3057. doi: 10.1200/JCO.24.00546. Epub 2024 Jun 25. PMID 38917371
- [Result] Diccianni MB, Kempinska K, Gangoti JA, Yu AL, Sorkin LS. Anti-GD2 induced allodynia in rats can be reduced by pretreatment with DFMO. PLoS One. 2020 Jul 22;15(7):e0236115. doi: 10.1371/journal.pone.0236115. eCollection 2020. PMID 32697811
- [Result] Salemi F, Alam W, Hassani MS, Hashemi SZ, Jafari AA, Mirmoeeni SMS, Arbab M, Mortazavizadeh SMR, Khan H. Neuroblastoma: Essential genetic pathways and current therapeutic options. Eur J Pharmacol. 2022 Jul 5;926:175030. doi: 10.1016/j.ejphar.2022.175030. Epub 2022 May 20. PMID 35605657
- [Result] Jabbari P, Hanaei S, Rezaei N. State of the art in immunotherapy of neuroblastoma. Immunotherapy. 2019 Jun;11(9):831-850. doi: 10.2217/imt-2019-0018. Epub 2019 May 16. PMID 31094257
- [Result] Pieniazek B, Cencelewicz K, Bzdziuch P, Mlynarczyk L, Lejman M, Zawitkowska J, Derwich K. Neuroblastoma-A Review of Combination Immunotherapy. Int J Mol Sci. 2024 Jul 15;25(14):7730. doi: 10.3390/ijms25147730. PMID 39062971
- [Result] Pinto NR, Applebaum MA, Volchenboum SL, Matthay KK, London WB, Ambros PF, Nakagawara A, Berthold F, Schleiermacher G, Park JR, Valteau-Couanet D, Pearson AD, Cohn SL. Advances in Risk Classification and Treatment Strategies for Neuroblastoma. J Clin Oncol. 2015 Sep 20;33(27):3008-17. doi: 10.1200/JCO.2014.59.4648. Epub 2015 Aug 24. PMID 26304901
- [Result] Newman EA, Abdessalam S, Aldrink JH, Austin M, Heaton TE, Bruny J, Ehrlich P, Dasgupta R, Baertschiger RM, Lautz TB, Rhee DS, Langham MR Jr, Malek MM, Meyers RL, Nathan JD, Weil BR, Polites S, Madonna MB; APSA Cancer committee. Update on neuroblastoma. J Pediatr Surg. 2019 Mar;54(3):383-389. doi: 10.1016/j.jpedsurg.2018.09.004. Epub 2018 Sep 19. PMID 30305231
- [Result] Hubbard AK, Spector LG, Fortuna G, Marcotte EL, Poynter JN. Trends in International Incidence of Pediatric Cancers in Children Under 5 Years of Age: 1988-2012. JNCI Cancer Spectr. 2019 Mar;3(1):pkz007. doi: 10.1093/jncics/pkz007. Epub 2019 Apr 9. PMID 30984908